CLINICAL TRIAL: NCT03035604
Title: Malnutrition in Older Cancer Patients
Brief Title: Comprehensive Nutritional Geriatric Assessments in Identifying Malnutrition in Older Cancer Participants
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0705; NCI-2018-01280 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0705 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nutritional geriatric assessment: Participants undergo nutritional geriatric assessment over 15 minutes in person or on the phone every 3 months for 12 months.
  Interventions: Other: Comprehensive Geriatric Assessment

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — Undergo nutritional geriatric assessment

SUMMARY:
This trial studies how well comprehensive nutritional geriatric assessments work in identifying malnutrition in older cancer participants. Comprehensive nutritional geriatric assessments may help doctors learn about ways to check for malnutrition (loss of weight/appetite that may result in health problems) that is due to cancer or cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether nutritional status, as determined by each of 4 screening tools (Mini Nutritional Assessment [MNA], weight loss, body mass index [BMI], and lean muscle mass), correlates with 6-month and 12-month mortality in older cancer patients after geriatric assessment, after adjusting for covariates.

II. To evaluate whether nutritional status, as determined by each of by 4 screening tools (MNA, weight loss, BMI, and lean muscle mass) correlates with 6-month and 12-month unplanned hospitalization in older cancer patients who undergo geriatric assessment, after adjusting for covariates.

III. To evaluate whether nutritional status, as determined by each of 4 screening tools (MNA, weight loss, BMI, and lean muscle mass) correlates with 6-month and 12-month hospital readmissions in older cancer patients who undergo geriatric assessment, after adjusting for covariates.

OUTLINE:

Participants undergo nutritional geriatric assessment over 15 minutes in person or on the phone every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* With hematologic and solid tumor cancers.
* Undergo a comprehensive geriatric assessment by a geriatrician.

Exclusion Criteria:

* Unable or unwilling to sign consent form.
* Life expectancy under 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants with hematologic and solid tumor cancers, undergo a comprehensive geriatric assessment by a geriatrician
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | At 6 months
  The association between nutrition status and mortality (6-month and 1-year mortality since geriatric assessment) will be assessed by logistic regression analysis, considering mortality as a response variable. Univariate logistic regression analysis will be used to estimate the crude odds ratio, and multivariable logistic regression will be used to estimate the adjusted odds ratio, after controlling for potential confounder variables, such as age, race, cancer type, cancer stage, co-morbidity, cognitive status), and frailty. ROC curve to predict 6-month and 1-year mortality will be constructed for nutritional status, as determined by each screening tool. The area under the ROC curve, sensitivity, and specificity and 95% confidence intervals will be obtained for each screening tool.

SECONDARY OUTCOMES:
Mortality | At 1 year
  The association between nutrition status and mortality (6-month and 1-year mortality since geriatric assessment) will be assessed by logistic regression analysis, considering mortality as a response variable. Univariate logistic regression analysis will be used to estimate the crude odds ratio, and multivariable logistic regression will be used to estimate the adjusted odds ratio, after controlling for potential confounder variables, such as age, race, cancer type, cancer stage, co-morbidity, cognitive status), and frailty. ROC curve to predict 6-month and 1-year mortality will be constructed for nutritional status, as determined by each screening tool. The area under the ROC curve, sensitivity, and specificity and 95% confidence intervals will be obtained for each screening tool.
Unplanned hospitalization rate | At 6 months and 1 year
  The associations between nutrition status and unplanned hospitalization will be assessed by logistic regression analysis. Univariate logistic regression analysis will be used to get the crude odds ratio, and multivariable logistic regression will be used to get the adjusted odds ratio, after controlling for potential confounder variables, such as age, race, cancer type, cancer stage, co-morbidity, cognitive status, and frailty. Patients who died before 6 months or 1 year from geriatric test will be considered as having unplanned 6-month or 1-year hospitalization. ROC curve to predict each of secondary outcomes will be constructed for nutritional status, as determined by each screening tool. The area under the ROC curve, sensitivity, and specificity and 95% confidence intervals will be obtained for each screening tool. Descriptive statistics will be used to summarize data. Two sample t-test or Wilcoxon rank-sum test will be used for the comparison in numeric variables.
Hospital readmission rate | At 6 months
  The associations between nutrition status and hospital readmissions will be assessed by logistic regression analysis. Univariate logistic regression analysis will be used to get the crude odds ratio, and multivariable logistic regression will be used to get the adjusted odds ratio, after controlling for potential confounder variables, such as age, race, cancer type, cancer stage, co-morbidity, cognitive status, and frailty. Patients who died before 6 months or 1 year from geriatric test will be considered as having unplanned 6-month or 1-year hospitalization. ROC curve to predict each of secondary outcomes will be constructed for nutritional status, as determined by each screening tool. The area under the ROC curve, sensitivity, and specificity and 95% confidence intervals will be obtained for each screening tool. Descriptive statistics will be used to summarize data. Two sample t-test or Wilcoxon rank-sum test will be used for the comparison in numeric variables.
Re-hospitalization rate | At 1 year
  The associations between nutrition status and hospital readmissions will be assessed by logistic regression analysis. Univariate logistic regression analysis will be used to get the crude odds ratio, and multivariable logistic regression will be used to get the adjusted odds ratio, after controlling for potential confounder variables, such as age, race, cancer type, cancer stage, co-morbidity, cognitive status, and frailty. Patients who died before 6 months or 1 year from geriatric test will be considered as having unplanned 6-month or 1-year hospitalization. ROC curve to predict each of secondary outcomes will be constructed for nutritional status, as determined by each screening tool. The area under the ROC curve, sensitivity, and specificity and 95% confidence intervals will be obtained for each screening tool. Descriptive statistics will be used to summarize data. Two sample t-test or Wilcoxon rank-sum test will be used for the comparison in numeric variables.

CONTACTS AND LOCATIONS:
Overall Officials: Mehnaz Shafi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org